CLINICAL TRIAL: NCT01045876
Title: The Effect of Dexamethasone on Plasma Cortisol Levels, Pain and PONV in Female Patients Undergoing Thyroid Surgery
Brief Title: The Effect of Dexamethasone on Cortisol Levels in Patients Undergoing Thyroid Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of resources
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Jill Osborn, Anesthesiologist, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SPH-1515-DA
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Adrenal Insufficiency
Keywords: Randomized controlled trial; Dexamethasone; Single dose; Preoperative; Plasma Cortisol level
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — One dose of 8 mg of Dexamethasone intravenously at induction of anesthesia
  Arms: Dexamethasone
Other: Placebo — 2 ml of 0.9% Saline Solution administered intravenously at induction of anesthesia
  Arms: Placebo

SUMMARY:
Many drugs are used to prevent nausea and vomiting and pain after surgery. In this study the investigators will be looking at a drug, dexamethasone, which is commonly used to prevent nausea and vomiting and pain after surgery but has other side effects. Dexamethasone is a man-made drug that is commonly used during surgery but also can affect naturally occuring hormones. In this study the investigators will be looking at dexamethasone's effect on a number of naturally occuring hormones over a twenty four hour period after thyroid surgery. The investigators hypothesize that plasma cortisol levels will be decreased following administration of dexamethasone.

DETAILED DESCRIPTION:
Purpose To examine the effect of dexamethasone, on plasma cortisol levels, postoperative pain, nausea and vomiting in patients undergoing thyroid surgery.

Hypothesis That dexamethasone administered at induction of anesthesia will result in reduced plasma cortisol levels, postoperative pain, nausea and vomiting.

Justification Dexamethasone is a synthetic steroid medication used routinely to prevent nausea and vomiting in patients undergoing general anesthetic. Administration of exogenous steroids can suppress production of endogenous steroids including cortisol.

Currently, no data exists describing the degree of suppression of cortisol production by a single preoperative dose of dexamethasone. This information would guide physicians prescribing dexamethasone in the perioperative period.

Objectives To compare plasma cortisol levels in patients receiving dexamethasone versus placebo at induction of anesthesia. To investigate the effect of dexamethasone on postoperative pain, nausea and vomiting.

Research Methods A prospective, randomized, controlled, double-blinded study conducted at a single center. Thirty patients will be recruited and randomly assigned to dexamethasone or placebo groups, in accordance with sample size calculations. A placebo group is necessary to eliminate the effects of potential confounding factors.

Statistical Analysis An interim analysis will be conducted to confirm the sample size calculation. Plasma cortisol level will be analyzed using 2-way analysis of variance (ANOVA). Secondary outcome measures will be analyzed with appropriate parametric or nonparametric methods.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients
* Undergoing thyroid surgery
* Euthyroid patients
* Qualify as Class I or II according to the American Society of Anesthesiologists physical status classification system
* Written informed consent

Exclusion Criteria:

* Patients who have medical conditions associated with abnormalities of the hypothalamic-pituitary-adrenal axis which might alter plasma cortisol levels will be excluded from the study. This category includes the following conditions:

  1. A diagnosis of anxiety, depression or bipolar disorder
  2. Disorders of the central nervous system, pituitary gland or hypothalamic-pituitary-adrenal axis
  3. Diabetes mellitus
  4. Pathological conditions affecting cortisol metabolism, including liver disease
  5. Chronic renal failure
  6. Alcoholism
  7. Obesity
  8. Anorexia nervosa/ starvation
  9. High estrogen states, including pregnancy or use of OCP
* Patients taking medication which might alter the normal function of the hypothalamic-pituitary-adrenal axis. This category includes:

  1. Patients taking exogenous steroid medication which would suppress normal cortisol production.
  2. Patients taking medication which alters steroid metabolism, including barbiturates, phenytoin and rifampicin.
* Patients who have a known history of allergy, sensitivity or any other form of reaction to dexamethasone will be excluded from this study as they would be at risk of further reaction to dexamethasone.
* Patients who have previously been included in this study will be excluded from further recruitment.
* Patients who will undergo lateral neck dissection in association with the thyroid surgery will be excluded from the study as they will experience greater pain levels.
* Patients who participate in other clinical studies during this study or in the 14 days prior to admission to this study will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2014-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Plasma Cortisol level. | One, eight and twenty-four hours following Dexamethasone administration.

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting. | Twenty-four hours following surgery.
Pain intensity measured on the visual analogue scale. | Twenty-four hours following surgery
Plasma Estradiol level. | One, eight and twenty-four hours following dexamethasone administration.
Plasma Progesterone level. | One, eight and twenty-four hours following dexamethasone administration
Plasma ACTH level | One, eight and twenty-four hours following dexamethasone administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Osborn, MD, Principal Investigator — St Paul's Hospital, Vancouver and University of British Columbia
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada